CLINICAL TRIAL: NCT04553029
Title: A Cross-sectional Survey Evaluating Prevalence, Severity and Associated Factors in East Asian Women With Moderate To-severe Menopause-related Vasomotor Symptoms (MR-VMS)
Brief Title: A Survey Evaluating Prevalence, Severity and Associated Factors in East Asian Women With Moderate-to-severe Menopause-related Vasomotor Symptoms (MR-VMS)
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Singapore Pte. Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 2693-MA-3289
Record Dates: First submitted 2020-09-14; First posted 2020-09-17 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2020-11

CONDITIONS: Menopause
Keywords: peri-menopausal; hormone replacement therapy; menopause; VMS; post-menopausal; menopausal; Vasomotor Symptoms; HRT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Peri-menopausal woman: Grouping is based on Peri-menopausal woman
  Interventions: Other: No intervention
- Group 2: Post- menopausal woman: Grouping is based on Post-menopausal woman
  Interventions: Other: No intervention
- Group 3: Peri-menopausal woman: moderate-to-severe MR-VMS: Grouping is based on Peri-menopausal woman with moderate-to-severe vasomotor symptoms (MR-VMS)
  Interventions: Other: No intervention
- Group 4: Post-menopausal woman: moderate-to-severe MR-VMS: Grouping is based on Post-menopausal woman with moderate-to-severe vasomotor symptoms (MR-VMS)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a cross-sectional survey study evaluating prevalence, severity and associated factors in women with moderate-to-severe menopause-related vasomotor symptoms (MR-VMS).

SUMMARY:
The purpose of this study is to estimate the prevalence of Vasomotor Symptoms (VMS) and prevalence of moderate to severe VMS in peri-menopausal women and post-menopausal women aged 40-65 in East Asia (China, South Korea and Taiwan) and the proportion of the following subpopulations: Hormone Replacement Therapy (HRT)-eligible and willing to take HRT; HRT-eligible and HRT-averse (i.e. not willing to take HRT); HRT-ineligible due to contra-indications/high-risk; and HRT-stoppers.

The study will also assess Health Related Quality of Life (HRQoL) and VMS related productivity loss among perimenopausal and post-menopausal women with moderate-to-severe MR-VMS and the respondents' attitudes toward prescription treatments.

DETAILED DESCRIPTION:
The study will recruit women of 40-65 years old from an established consumer panel in China, South Korea, and Taiwan.

Women who meet the inclusion criteria for Part I will be recruited to sign the informed consent form (ICF) and participate in Part I of the survey.

Based on the information collected in Part I of the survey, peri- and post-menopausal women who meet the inclusion criteria for Part II will be directed to Part II of the survey. The survey will be terminated for women who do not meet the inclusion criteria for Part II.

ELIGIBILITY:
Inclusion Criteria (part I):

* Evidence of peri-menopause (changes in the regular period in terms of irregularity in the length of the period, the time between periods, and the level of flow), or
* Evidence of post-menopause (spontaneous amenorrhea over 12 months)

Inclusion Criteria (part II):

* Presence of moderate-to-severe menopause-related vasomotor symptoms (MR-VMS); Moderate: sensation of heat with sweating, able to continue activity; Severe: sensation of heat with sweating, causing cessation of activity)

Exclusion Criteria (part I):

* No evidence of peri-menopause or post-menopause, or
* Women who are currently participating or have participated in menopause-related vasomotor symptoms (MR-VMS) clinical trials

Exclusion Criteria (part II):

* Subjects who are treated with tamoxifen, aromatase inhibitors or Gonadotropin-releasing hormone (GnRH) agonists/antagonists for cancer or any other medical condition, or
* Subjects who have mild menopause-related vasomotor symptoms (MR-VMS) only

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: peri-menopausal women and post-menopausal women aged 40-65 in East Asia (China, South Korea and Taiwan)
Sampling Method: Probability Sample
Enrollment: 3399 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Prevalence of Vasomotor Symptoms (VMS) in peri-menopausal women and post-menopausal women aged 40-65 | 1 day (once through survey)
  Prevalence of VMS in peri-menopausal women and post-menopausal women aged 40-65. Peri-menopause is defined as changes in the regular period in terms of irregularity in the length of the period, the time between periods, and the level of flow. Post-menopause is defined as spontaneous amenorrhea over 12 months.
Prevalence of moderate-to-severe Vasomotor Symptoms (VMS) in peri-menopausal women and post-menopausal women aged 40-65 | 1 day (once through survey)
  Prevalence of moderate-to-severe Vasomotor Symptoms (VMS) cases in peri-menopausal women and post-menopausal women aged 40-65 will be evaluated.
Severity of Vasomotor Symptoms (VMS) symptoms based on pre-defined definitions for severity among peri-menopausal women and post-menopausal women aged 40-65 | 1 day (once through survey)
  Severity of Vasomotor Symptoms (VMS) in peri-menopausal women and post-menopausal women aged 40-65 will be evaluated following the Food and Drug Administration (FDA) Guidelines. The severity of VMS symptoms may range from: absence of symptoms (no sensation of heat or sweating), mild (the sensation of feeling hot without sweating), moderate (the sensation of feeling hot, accompanied by sweating, and able to maintain activity), and severe (the sensation of feeling hot, accompanied by sweating, and needing to cease activity).
Proportion of participants Hormone Replacement Therapy (HRT) eligible and willing to take HRT | 1 day (once through survey)
  Number of participants eligible and willing to take Hormone Replacement Therapy (HRT) compared to number of participants evaluated.
Proportion of participants Hormone Replacement Therapy (HRT) eligible and HRT averse | 1 day (once through survey)
  Number of participants eligible and not willing to take Hormone Replacement Therapy (HRT) compared to number of participants evaluated.
Proportion of participants Hormone Replacement Therapy (HRT) ineligible due to contra-indications/high risk | 1 day (once through survey)
  Number of participants ineligible to take Hormone Replacement Therapy (HRT) due to contra-indications/high risk compared to number of participants evaluated.
Proportion of participants that stopped Hormone Replacement Therapy (HRT) | 1 day (once through survey)
  Number of participants that stopped Hormone Replacement Therapy (HRT) compared to number of participants evaluated.

SECONDARY OUTCOMES:
Health Related Quality of Life (HRQoL) measured by Menopause Specific Quality of Life Questionnaire (MENQOL) | 1 day (once through survey)
  The Menopause Specific Quality of Life Questionnaire (MENQOL) measures the overall score and four domain-specific scores assessing wellbeing (Vasomotor; Psychosocial; Physical; Sexual). Scores range from 1-8 with a higher score indicating worsening/increasing bothersomeness by the symptom experience. The MENQOL recall period is 7 days prior to survey.
Health Related Quality of Life (HRQoL) measured by Work Productivity and Activity Impairment (WPAI) | 1 day (once through survey)
  The Work Productivity and Activity Impairment (WPAI) measures Four domain specific scores assessing work productivity and activity impairment over the previous week (Absenteeism; Presenteeism; Mean work productivity; Activity impairment). Scores range from 0 to 100%. The four scores were expressed as impairment percentages with a higher score indicating less productivity and greater activity impairment. The WPAI recall period is 7 days prior to survey.
Health Related Quality of Life (HRQoL) measured by Treatment history related to menopause-related vasomotor symptoms (MR-VMS) | 1 day (once through survey)
  Menopause-related vasomotor symptoms (MR-VMS) treatment history will be evaluated by Hospital/clinics visiting history related to MR-VMS; past treatments and current treatments (e.g., hormone therapy, antidepressants, herbal medicine, acupuncture).
Health Related Quality of Life (HRQoL) measured by Patient attitudes towards prescription treatment choices in participants with moderate-to-severe MR-VMS | 1 day (once through survey)
  Patient attitudes towards prescription treatment choices will be evaluated using the following reasons/ factors: Reasons for seeking /not seeking treatments; Reasons for visiting/not visiting hospital/clinics; Awareness of long-term health risks if remain untreated; Willingness to seek for care/treatment if patients were aware of long-term health risks associated with leaving moderate-to-severe MR-VMS untreated; Reasons for choosing the current prescription treatments; Reasons for discontinuation of the previous prescription treatment; Factors determining prescription treatment choices and preference (for those who are not currently receiving treatment); Willingness toward new pharmacologic treatments; Key concerns of new pharmacologic treatments (for those who are not willing to try new treatment); and Key expectations of new pharmacologic treatments (for those willing to try new treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Astellas Pharma Singapore Pte. Ltd.
Locations (3):
- Site CN86002, Beijing, China
- Site KR82001, Seoul, South Korea
- Site TW88601, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.